CLINICAL TRIAL: NCT00884832
Title: A Placebo-Controlled Study of Clonidine for Fecal Incontinence.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, Adil Bharucha, PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 08-005892; R01DK078924 (NIH); UL1RR024150 (NIH)
Record Dates: First submitted 2009-04-17; First posted 2009-04-21 (Estimated); Results first posted 2014-03-06 (Estimated); Last update posted 2014-03-06 (Estimated); Status verified 2014-01

CONDITIONS: Fecal Incontinence
Keywords: fecal incontinence; stool leakage; incontinence; FI; Urge predominant fecal incontinence
MeSH Terms: conditions — Fecal Incontinence | interventions — Clonidine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral Clonidine (Experimental): Subjects randomized to Clonidine will take 0.1 mg of the medication orally twice a day for a total of 4 weeks.
  Interventions: Drug: Clonidine
- Oral Placebo (Placebo Comparator): Subjects randomized to the placebo group will also take 0.1 mg of matching placebo pills orally twice a day for a total of 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clonidine — Subjects randomized to Clonidine will take 0.1 mg of the medication orally twice a day for a total of 4 weeks.
  Other Names: Kapvay; Nexiclon; Catapres
  Arms: Oral Clonidine
Drug: Placebo — Subjects randomized to the placebo group will also take 0.1 mg of matching placebo pills orally twice a day for a total of 4 weeks.
  Arms: Oral Placebo

SUMMARY:
Fecal incontinence is the involuntary leakage of stool from the anus. Doctors at Mayo Clinic are doing a research study to assess the effects of a medication, clonidine, on fecal incontinence and rectal functions in women. Clonidine has been approved by the Food and Drug Administration (FDA) for treating high blood pressure, but not for treating incontinence and rectal functions. The hypothesis of this study is clonidine will improve fecal incontinence, increase rectal capacity and reduce rectal sensation to a greater extent than placebo in women.

DETAILED DESCRIPTION:
Available therapeutic options for idiopathic fecal incontinence (FI) are limited and unsatisfactory. In addition to weak anal sphincters, our data suggest that reduced rectal capacity may contribute to rectal hypersensitivity and the symptom of rectal urgency in FI. During a 4 week study, oral clonidine restored rectal capacity and improved fecal continence in women with urge-predominant FI. Clonidine improves fecal continence and stool consistency in diarrhea-predominant irritable bowel syndrome (IBS). Therefore, we now propose a placebo-controlled study of clonidine for FI. Our aims are to (i) compare the effects of clonidine and placebo, to be given for 4 weeks, on symptoms, anal pressures, rectal compliance and sensation in women with FI. Forty four women (18-75 y) with urge predominant "idiopathic" FI and ≥ 4 episodes of FI during a 4 week screening period will be recruited to this study. Thereafter, patients will be treated with clonidine or placebo for 4 weeks. Bowel symptoms will be recorded in a diary. Anal sphincter pressures, rectal compliance and sensation will be evaluated before and during treatment with clonidine.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-75 years with urge predominant FI, as defined by a validated questionnaire, for greater than or equal to 1 year duration will be eligible to participate
* Absence of organic disease (i.e., ulcerative colitis, cancer) as evidenced by colonoscopy, or barium enema and sigmoidoscopy within the last 3 years

Exclusion Criteria:

* History of clinically significant cardiovascular or pulmonary disease or EKG abnormalities within the last 6 months [i.e., atrial flutter or fibrillation, sinus tachycardia (> 110/minute) or bradycardia (< 45 beats/minute), or prolonged corrected QT (QTc) interval (> 460 msec)
* Current or past history of rectal cancer, scleroderma, inflammatory bowel disease, congenital anorectal abnormalities, greater than or equal to Grade 2 rectal prolapse, history of rectal resection or pelvic irradiation
* Neurological disorders - Spinal cord injuries, dementia (Mini-mental status score <20/25), multiple sclerosis, Parkinson's disease, peripheral neuropathy
* Conditions precluding safe use of clonidine, i.e., symptomatic hypotension, or systolic blood pressure of <100 mm Hg on initial screening visit
* Pregnant or nursing women
* Severe diarrhea during the run in phase defined as greater than 6 liquid stools daily (Bristol 6 or 7)
* Medications: Absolute - opioid analgesics, anticholinergic drugs [low doses of tricyclic antidepressants, e.g., nortriptyline (up to 50 mg/day) or amitriptyline (up to 25 mg/day) will be permitted provided they were begun 3 months prior to the screening period]
* Medications: Relative - other antihypertensive agents (i.e., if there is concern about synergistic effects and hypotension)

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2008-10; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adil E Bharucha, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Bharucha AE, Fletcher JG, Camilleri M, Edge J, Carlson P, Zinsmeister AR. Effects of clonidine in women with fecal incontinence. Clin Gastroenterol Hepatol. 2014 May;12(5):843-851.e2; quiz e44. doi: 10.1016/j.cgh.2013.06.035. Epub 2013 Jul 23. PMID 23891925

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted between January 2009 and April 2012.
Period: Overall Study
Arm/Group | Oral Clonidine | Oral Placebo
Started | 22 | 22
Completed | 22 | 21
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Clonidine | Oral Placebo | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (10.88) | 57 (11.86) | 57.38 (11.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 22 | 44
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 22 | 22 | 44
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 30.3 (1.09) | 28.0 (6.35) | 29.14 (5.81)
Hysterectomy [Number; unit: participants] — Number of participants who had previously had a hysterectomy at baseline.
  participants
    Hysterectomy | 9 | 11 | 20
    No Hysterectomy | 13 | 11 | 24
Functional diarrhea or Diarrhea-predominant Irritable Bowel Syndrome (IBS) [Number; unit: participants]
  Subjects with diarrhea | 9 | 13 | 22
  Subjects without diarrhea | 13 | 9 | 22

OUTCOME MEASURES:

1. Primary Outcome: Mean Fecal Incontinence and Constipation Assessment (FICA) Score
Description: The FICA severity scale has 4 items (frequency, type, amount of leakage, and presence of urgency) and is used to rate the severity of fecal incontinence. The parameter was computed from values in the weekly diaries. The FICA score can range from 1 to 13. Symptom severity scores of 1-6, 7-10, and 11-13 are categorized as mild, moderate, and severe, respectively. Scores were averaged over the 4 week baseline period and the 4 week treatment periods.
Time Frame: 4 weeks baseline, 4 weeks treatment
Population: Intent to treat analysis
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Oral Clonidine | Oral Placebo
Number analyzed (Participants) | 22 | 22
units on a scale
  4 weeks baseline | 8.1 (0.4) | 9.1 (0.3)
  4 weeks treatment | 6.5 (0.6) | 7.6 (0.5)

2. Secondary Outcome: Mean Number of Days With Fecal Incontinence
Description: Values were averaged over 4 week baseline and 4 week treatment periods.
Time Frame: 4 weeks baseline, 4 weeks treatment
Population: Intent to treat analysis
Measure: Mean (Standard Error); unit: days
Arm/Group | Oral Clonidine | Oral Placebo
Number analyzed (Participants) | 22 | 22
days
  4 weeks baseline | 13 (1) | 16 (2)
  4 weeks treatment | 8 (1) | 11 (2)

3. Secondary Outcome: Mean Number of Fecal Incontinence Episodes
Description: Values were averaged over 4 week baseline and 4 week treatment periods.
Time Frame: 4 weeks baseline, 4 weeks treatment
Population: Intent to treat analysis
Measure: Mean (Standard Error); unit: number of episodes
Arm/Group | Oral Clonidine | Oral Placebo
Number analyzed (Participants) | 22 | 22
number of episodes
  4 weeks baseline | 20 (3) | 31 (5)
  4 weeks treatment | 12 (3) | 19 (4)

4. Secondary Outcome: Mean Percentage of Bowel Movements Which Were Incontinent
Description: Values were averaged over 4 week baseline and 4 week treatment periods.
Time Frame: 4 weeks baseline, 4 weeks treatment
Population: Intent to treat analysis
Measure: Mean (Standard Error); unit: percentage of bowel movements
Arm/Group | Oral Clonidine | Oral Placebo
Number analyzed (Participants) | 22 | 22
percentage of bowel movements
  4 weeks baseline | 31 (4) | 40 (6)
  4 weeks treatment | 24 (5) | 27 (6)

5. Secondary Outcome: Mean Severity of Fecal Incontinence
Description: The Fecal Incontinence Severity Index was used to compute the severity of fecal incontinence (FI). It is a validated 4-item scale used to assess the frequency of 4 different types of FI (gas, mucus, liquid stool, solid stool). The subject responses are weighted and summed for the 4 types of FI. Scores could range from 0 (no symptoms) to 61 (very frequent FI). Values were computed from pre- and post- treatment questionnaires.
Time Frame: 4 weeks baseline, 4 weeks treatment
Population: Intent to treat analysis
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Oral Clonidine | Oral Placebo
Number analyzed (Participants) | 22 | 22
units on a scale
  4 weeks baseline | 36.2 (2.7) | 37.3 (2.5)
  4 weeks treatment | 29.3 (2.8) | 31.2 (2.7)

6. Secondary Outcome: Impact of Fecal Incontinence on Baseline Quality of Life
Description: Scores were computed from a pre-treatment questionnaire, the Fecal Incontinence Quality of Life Scale. This scale is composed of a total of 29 items; these items form four scales: Lifestyle (10 items) Coping/Behavior (9 items), Depression/Self Perception (7 items), and Embarrassment (3 items).
  Scales range from 1 to 4; with a 1 indicating a lower functional status of quality of life. Scales scores are the average (mean) response to all items in the scale (that is, add the responses to all questions in a scale together and then divide by the number of items in the scale, adjusting for missing values).
Time Frame: 4 weeks baseline
Population: Intent to treat analysis
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Oral Clonidine | Oral Placebo
Number analyzed (Participants) | 22 | 22
units on a scale
  Lifestyle score | 2.8 (0.2) | 2.3 (0.2)
  Coping score | 1.8 (0.1) | 1.6 (0.1)
  Depression score | 3.2 (0.2) | 2.9 (0.2)
  Embarrassment score | 2.2 (0.2) | 2.3 (0.2)

7. Secondary Outcome: Impact of Fecal Incontinence on Post-Treatment Quality of Life
Description: Scores were computed from a post-treatment questionnaire, the Fecal Incontinence Quality of Life Scale. This scale is composed of a total of 29 items; these items form four scales: Lifestyle (10 items) Coping/Behavior (9 items), Depression/Self Perception (7 items), and Embarrassment (3 items).
  Scales range from 1 to 4; with a 1 indicating a lower functional status of quality of life. Scales scores are the average (mean) response to all items in the scale (that is, add the responses to all questions in a scale together and then divide by the number of items in the scale, adjusting for missing values).
Time Frame: after 4 weeks treatment
Population: Intent to treat analysis
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Oral Clonidine | Oral Placebo
Number analyzed (Participants) | 22 | 22
units on a scale
  Lifestyle score | 3.1 (0.2) | 2.7 (0.2)
  Coping score | 2.3 (0.2) | 2.1 (0.1)
  Depression score | 3.5 (0.1) | 3.2 (0.2)
  Embarrassment score | 2.8 (0.2) | 2.5 (0.2)

8. Secondary Outcome: Satisfaction With Treatment
Description: This parameter was determined by a 100 mm visual analog scale, with possible scores ranging from 0 = "Not satisfied at all (no relief of symptoms)" to 100 = "Completely satisfied (symptoms resolved)." The parameter was computed from weekly diaries. Scores were averaged over the 4 week baseline period and the 4 week treatment periods.
Time Frame: 4 weeks baseline, 4 week treatment
Population: Intent to treat analysis
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Oral Clonidine | Oral Placebo
Number analyzed (Participants) | 22 | 22
units on a scale
  4 weeks baseline | 22 (6) | 18 (4)
  4 weeks treatment | 47 (6) | 38 (6)

9. Secondary Outcome: Percentage of Bowel Movements Preceded by Rectal Urgency
Description: Rectal urgency is defined as a sudden, irresistible need to have a bowel movement. Scores were averaged over the 4 week baseline period and the 4 week treatment periods.
Time Frame: 4 weeks baseline, 4 weeks treatment
Population: Intent to treat analysis
Measure: Mean (Standard Error); unit: percentage of bowel movements
Arm/Group | Oral Clonidine | Oral Placebo
Number analyzed (Participants) | 22 | 22
percentage of bowel movements
  4 weeks baseline | 55 (4) | 59 (5)
  4 weeks treatment | 46 (6) | 46 (6)

10. Secondary Outcome: Percentage of Bowel Movements With Semi-formed and Loose Stools in Subjects With and Without Diarrhea
Description: The percentage of bowel movements with semi-formed and loose stools was defined as those with a score of 5-7 on the Bristol stool form scale.
Time Frame: 4 weeks baseline, 4 weeks treatment
Population: Intent to treat analysis
Measure: Mean (Standard Error); unit: percentage of bowel movements
Arm/Group | Oral Clonidine | Oral Placebo
Number analyzed (Participants) | 22 | 22
percentage of bowel movements
  4 weeks baseline, subjects without diarrhea | 19.4 (4.9) | 25.5 (6.2)
  4 weeks baseline, subjects with diarrhea | 47.5 (8.1) | 51.6 (6.4)
  4 weeks treatment, subjects without diarrhea | 14 (4.2) | 16 (7.2)
  4 weeks treatment, subjects with diarrhea | 31.2 (7) | 49 (5.5)
Statistical Analysis 1: Comparison: Oral Clonidine vs Oral Placebo; Proportion of semi-formed and loose stools (Bristol Form 5-7) associated with diarrhea subgroup versus no diarrhea subgroup; Test type: Superiority or Other; p < 0.001, ANCOVA

11. Secondary Outcome: Percentage of Bowel Movements With Semi-formed and Loose Stools Post-treatment Adjusted for Baseline
Description: The percentage of bowel movements with semi-formed and loose stools was defined as those with a score of 5-7 on the Bristol stool form scale. The "adjustment for baseline" was an analysis of covariance (ANCOVA) where the covariate was the baseline version of the endpoint.
Time Frame: 4 weeks treatment
Population: Intent to treat analysis
Measure: Mean (Standard Error); unit: percentage of bowel movements
Arm/Group | Oral Clonidine | Oral Placebo
Number analyzed (Participants) | 22 | 22
percentage of bowel movements
  Subjects with diarrhea | 23.6 (4.8) | 38.7 (4.3)
  Subjects without diarrhea | 25.4 (4.3) | 22.8 (4.8)
Statistical Analysis 1: Comparison: Oral Clonidine vs Oral Placebo; Test type: Superiority or Other; p = 0.018, ANCOVA
Statistical Analysis 2: Comparison: Oral Clonidine vs Oral Placebo; drug*group interactions; Test type: Superiority or Other; p = 0.047, ANCOVA

12. Secondary Outcome: Percentage of Days With Fecal Incontinence (FI)
Time Frame: 4 weeks baseline, 4 weeks treatment
Measure: Mean (Standard Error); unit: percentage of days
Arm/Group | Oral Clonidine | Oral Placebo
Number analyzed (Participants) | 22 | 22
percentage of days
  4 weeks baseline, subjects without diarrhea | 28.7 (5.5) | 37.8 (10.6)
  4 weeks baseline, subjects with diarrhea | 35.4 (7.2) | 42.1 (8.1)
  4 weeks treatment, subjects without diarrhea | 23.2 (7.1) | 18.7 (5.4)
  4 weeks treatment, subjects with diarrhea | 24.3 (8.5) | 33.3 (9.8)

13. Secondary Outcome: Percentage of Days With FI Post-treatment Adjusted for Baseline
Description: The "adjustment for baseline" was an analysis of covariance (ANCOVA) where the covariate was the baseline version of the endpoint.
Time Frame: 4 weeks treatment
Measure: Mean (Standard Error); unit: percentage of days
Arm/Group | Oral Clonidine | Oral Placebo
Number analyzed (Participants) | 22 | 22
percentage of days
  Subjects without diarrhea | 42.54 (5.92) | 31.42 (6.97)
  Subjects with diarrhea | 27.79 (6.97) | 39.51 (5.94)
Statistical Analysis 1: Comparison: Oral Clonidine vs Oral Placebo; Test type: Superiority or Other; p = 0.082, ANCOVA

ADVERSE EVENTS:
Arm/Group | Oral Clonidine | Oral Placebo
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 19/22 | 7/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Clonidine (N=22) | Oral Placebo (N=22)
Dry Mouth (Gastrointestinal disorders) | 16 (16) | 1 (1)
Drowsiness (General disorders) | 5 (5) | 3 (3)
Lightheadedness (General disorders) | 6 (6) | 2 (2)
Fatigue (General disorders) | 8 (8) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No